CLINICAL TRIAL: NCT00439283
Title: Study of Two Schedules of Infliximab Maintenance Therapy in Ankylosing Spondylitis: Comparison of Infusion Every 6 Weeks Versus Infusion on Demand
Brief Title: Study of Two Schedules of Infliximab Maintenance Therapy in Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association de Recherche Clinique en Rhumatologie (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A R C R 2003 - 01 / PO 3353
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; infliximab; Systematic regimen; On-demand regimen
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: infliximab
Drug: methotrexate

SUMMARY:
Continuous treatment with the anti-tumor necrosis factor alpha monoclonal antibody infliximab is efficacious in ankylosing spondylitis (AS), whereas treatment discontinuation results in disease relapse, with variable delay. Objective of this study was to compare efficacy between a continuous treatment with infliximab, and a treatment adapted to symptoms recurrence. Addition of methotrexate (MTX)to infliximab was also tested.

DETAILED DESCRIPTION:
Patients with active AS were randomly assigned to receive infliximab every 6 weeks (Q6), or only upon symptoms recurrence (on-demand), following a loading regimen of infusions at weeks 0, 2, and 6. Patients in the latter group were randomly assigned to receive MTX or not, starting 4 weeks prior to infliximab. Monitoring was performed over one year. The primary end point was the proportion of patients with a 20% improvement response according to the ASsessment in Ankylosing Spondylitis (ASAS) criteria, at week 54.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years old)
* With a diagnosis of AS
* With at least one of the following evidences for active inflammation, present within 3 months before inclusion: a serum C-reactive protein (CRP) level above twice the upper limit value of the normal range, a positive magnetic resonance imaging of the spine or sacro-iliac joints, a vascularized enthesitis by power-Doppler ultrasound technic.
* Presence of clinically active axial disease, as defined by 1) a Bath AS Disease Activity Index (BASDAI) (18) of ≥ 3/10, and 2) a score of ≥ 3/10 for axial pain (second item of BASDAI).
* Disease-modifying antirheumatic drugs (DMARDs), such as sulphasalazine, methotrexate, hydroxychloroquine, intra-muscular gold, thiol compound, cyclosporin, intravenous biphosphonate had to be discontinued for at least 4 weeks before inclusion.
* Dosages of NSAIDs and corticosteroid were required to remain stable for at least 4 weeks before inclusion.
* A negative pregnancy test result was required for non menopausal female patients, and contraception during the study period and for six months after the last infusion of infliximab was recommended to all patients of childbearing potential.

Exclusion Criteria:

* Pregnancy.
* Breastfeeding.
* Vaccination with a live organism during the last month.
* Present infection or any episode of serious infection within the last three months.
* Active malignancy within the previous five years.
* Alcohol or drug addiction.
* Severe chronic concomitant disease.
* Administration of an investigational drug within the last three months, or of any known TNF inhibitor therapy in the past (such as thalidomide, infliximab or etanercept).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2003-04; Study Completion 2004-12

PRIMARY OUTCOMES:
The primary end point was the proportion of patients with a 20% improvement response according to the ASAS criteria, at week 54.

SECONDARY OUTCOMES:
Achievement of the ASAS50 and ASAS70.
The proportion of patients who experienced a partial remission, according to ASAS definition.
Improvement in independent components of the ASAS response criteria.
BASDAI.
SF-36.
Schober test.
Finger to floor test.
Chest expansion score.
Occiput-to-wall measurements.
Acute-phase reactants (erythrocyte sedimentation rate and C-reactive protein level).
Number of infusions administered after the loading regimen.
Number of patients requiring an increase in the dose of infliximab.
The area under the curves (AUCs) of the BASDAI recorded on a weekly basis on automatic phone server, calculated from week 0 through week 54.
The area under the curves (AUCs) of the global pain scores recorded on a weekly basis on automatic phone server, calculated from week 0 through week 54.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime DOUGADOS, Professor, Study Director — ARCR
Locations (31):
- France (31):
  - CHU Amiens, Amiens
  - CHU Hôpital Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de la Cavale Blanche, Brest
  - CHU Côte de Nacre, Caen
  - Hôpital Gilles de Corbeil, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - Hôpital Général, Dijon
  - CHU A. Michallon, Grenoble
  - Groupe Hospitalier du Havre, Le Havre
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU Hôpital Roger Salengro, Lille
  - CHU Dupuytren, Limoges
  - Centre Hospitalier Saint Philibert, Lomme
  - CH St Joseph - St Luc, Lyon
  - Hôpital de la Conception, Marseille
  - Hôpital Lapeyronie, Montpellier
  - CHU l'Archet 1, Nice
  - Hôpital Porte Madeleine, Orléans
  - Hôpital de la Pitié, Paris
  - Hôpital Cochin, Paris
  - CHU de Poitiers, Poitiers
  - CHU - Hôpital Sud, Rennes
  - CHU - Hôpital de Bois Guillaume, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Hautepierre, Strasbourg
  - Hôpital de Purpan, Toulouse
  - CHU Hôpital Trousseau, Tours
  - CHU Nancy-Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Fautrel B, Benhamou M, Breban M, Roy C, Lenoir C, Trape G, Baleydier A, Ravaud P, Dougados M. Cost effectiveness of two therapeutic regimens of infliximab in ankylosing spondylitis: economic evaluation within a randomised controlled trial. Ann Rheum Dis. 2010 Feb;69(2):424-7. doi: 10.1136/ard.2008.103887. Epub 2009 Sep 9. PMID 19740900
- [Derived] Breban M, Ravaud P, Claudepierre P, Baron G, Henry YD, Hudry C, Euller-Ziegler L, Pham T, Solau-Gervais E, Chary-Valckenaere I, Marcelli C, Perdriger A, Le Loet X, Wendling D, Fautrel B, Fournie B, Combe B, Gaudin P, Jousse S, Mariette X, Baleydier A, Trape G, Dougados M; French Ankylosing Spondylitis Infliximab Network. Maintenance of infliximab treatment in ankylosing spondylitis: results of a one-year randomized controlled trial comparing systematic versus on-demand treatment. Arthritis Rheum. 2008 Jan;58(1):88-97. doi: 10.1002/art.23167. PMID 18163509